CLINICAL TRIAL: NCT06065566
Title: Effect of Parenteral Glutamine on Myocardial Injury and Inflammation Biomarkers in Patients Undergoing to Cardiac Surgery With and Without Cardiopulmonary Bypass
Brief Title: Effect of Parenteral Glutamine on Myocardial Injury and Inflammation Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R-2019-1001-079
Record Dates: First submitted 2020-01-10; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Insufficiency;Cardiac
Keywords: Cardiovascular surgery; Glutamine; Heart damage markers
MeSH Terms: conditions — Heart Failure | interventions — Glutamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: 1. Once the candidate patients undergo surgery for cardiac surgery with and without cardiopulmonary bypass, the inclusion criteria will be verified. Once their inclusion in the study has been accepted, the patient must sign their informed consent letter and will be randomly assigned by closed envelope, to a study group or to a control group. The patient's weight and height will be taken once he accepts inclusion in the study and the data collection notebook will be filled.
  A. Study group: patients undergoing cardiac surgery with and without cardiopulmonary bypass, who will receive the dipeptide L-alanyl-L-glutamine, at a dose of 0.4 g / kg of weight 6 hours before the surgical intervention.
  B. Control group: patients undergoing cardiac surgery with and without cardiopulmonary bypass, who will receive the placebo in the form of saline solution in a volume similar to the control 6 hours before the surgical intervention.
Who Masked: Care Provider
Masking Description: A third person, the cardiothoracic surgery floor nurse, will assign the patients to the study group or control group by means of a sealed envelope. Registration will be carried out by this single person until the final results are revealed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients on bypass with cardiopulmonary bypass +gluta (Experimental): Patients operated on bypass with cardiopulmonary bypass + glutamine
  Interventions: Dietary Supplement: L-alanyl-L-glutamine dipeptide
- Patients on bypass + cardiopulmonary bypass + glutamine (Placebo Comparator): Patients operated on bypass with cardiopulmonary bypass + glutamine
  Interventions: Other: Placebo
- patients without bypass + cardiopulmonary bypass +glutamine (Experimental): Patients operated without bypass with cardiopulmonary bypass + glutamine
  Interventions: Dietary Supplement: L-alanyl-L-glutamine dipeptide
- Patients without bypass + cardiopulmonary bypass +placebo (Placebo Comparator): Patients operated without bypass with cardiopulmonary bypass + placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-alanyl-L-glutamine dipeptide — 1. Once the candidate patients undergo surgery for cardiac surgery with and without cardiopulmonary bypass, the inclusion criteria will be verified. Once their inclusion in the study has been accepted, the patient must sign their informed consent letter and will be randomly assigned by closed envelope, to a study group or to a control group. The patient's weight and height will be taken once he accepts inclusion in the study and the data collection notebook will be filled.
  A. Study group: patients undergoing cardiac surgery with and without cardiopulmonary bypass, who will receive the dipeptide L-alanyl-L-glutamine, at a dose of 0.4 g / kg of weight 6 hours before the surgical intervention.
  Other Names: Glutamine
  Arms: Patients on bypass with cardiopulmonary bypass +gluta; patients without bypass + cardiopulmonary bypass +glutamine
Other: Placebo — 1. Once the candidate patients undergo surgery for cardiac surgery with and without cardiopulmonary bypass, the inclusion criteria will be verified. Once their inclusion in the study has been accepted, the patient must sign their informed consent letter and will be randomly assigned by closed envelope, to a study group or to a control group. The patient's weight and height will be taken once he accepts inclusion in the study and the data collection notebook will be filled.
  B. Control group: patients undergoing cardiac surgery with and without cardiopulmonary bypass, who will receive the placebo in the form of saline solution in a volume similar to the control 6 hours before the surgical intervention.
  Other Names: Saline solution
  Arms: Patients on bypass + cardiopulmonary bypass + glutamine; Patients without bypass + cardiopulmonary bypass +placebo

SUMMARY:
The effect of parenteral glutamine on the biomarkers of myocardial injury and inflammation in patients undergoing cardiac surgery with and without cardiopulmonary bypass (DCP) will be analyzed. Randomized controlled clinical trial, from October 2018 to February 2022. 124 patients: 14 patients with DCP and 14 patients without DCP, both + glutamine (L-alanyl-L-glutamine dipeptide, at a dose of 0.4 g / kg) 6 hours before surgery and 14 patients with PCD and 14 patients without PCD + placebo (saline) 6 hours before surgery. Blood samples will be taken to measure the level of TROP-I, CPK-MB, HSP-70, TNFa, IL6, IL10 and PCR 1 hour before the administration of Glutamine / Placebo, 1 hour before surgery, then at 1 , 12 and 24 hours after surgery.

DETAILED DESCRIPTION:
Introduction: Cardiac surgery is performed in order to improve function and decrease the incidence of cardiac events. The provision of different metabolic substrates before and during cardiac surgery can have beneficial effects, limiting the damage caused by ischemia / reperfusion (I / R) induced by this type of surgery with and without cardiopulmonary bypass, reflected in a better recovery and survive. Glutamine (GLN) is a non-essential amino acid should be a primary part of medical and nutritional therapy in severe patients, since the reduction of this is associated in various critical conditions including multiple trauma, sepsis or after major surgery. In cardiac patients, the concentration of intracellular GLN is always reduced regardless of the surgical technique used.

Objective: To analyze the effect of parenteral glutamine in the biomarkers of myocardial injury and inflammation in patients undergoing cardiac surgery with and without cardiopulmonary bypass.

Hypothesis: Supplementation with parenteral glutamine reduces the expression of biomarkers of myocardial injury and inflammation in patients undergoing cardiac surgery with and without cardiopulmonary bypass.

Material and methods: A randomized controlled clinical trial will be carried out according to the consort 2010 criteria, in a period from October 2018 to September 2020. A total of 124 patients will be included that will be randomized as follows: 14 patients with referral cardiopulmonary + Glutamine and 14 patients without cardiopulmonary bypass + Glutamine who will receive the dipeptide L-alanyl-L-glutamine, at a dose of 0.4 g / kg of weight 6 hours before surgery and 14 patients with cardiopulmonary bypass and 14 patients without bypass cardiopulmonary, who will receive placebo in the form of saline solution in a volume similar to the control 6 hours before the surgical intervention. Blood samples will be taken to measure the level of TROP-I, CPK-MB, HSP-70, TNFα, IL6, IL10 and PCR 1 hour before the administration of Glutamine / Placebo, 1 hour before surgery, then 1 hour after of surgery and at 12 and 24 hours after surgery to be taken to the laboratory of the Post-surgical Coronary Care Unit and obtain the reading of the samples.

Statistical analysis: Averages and standard deviations for quantitative variables will be calculated; frequencies and proportions in qualitative variables. For statistical inference. Quantitative variables will be analyzed with Student's t-test for independent samples. ANOVA will be used for repeated measurements in each group to obtain the difference of the final value minus the initial one in the dependent variable (δ). Considering two-tailed tests, any value of p <0.05 will be considered statistically significant. The data will be captured in an Excel file and the statistical analysis will be carried out with the statistical package SPSS version 20.0, (SPSS, Chicago, ILL, U.S.A.).

Ethical considerations: This study will adhere to the principles emanating from the 18th medical assembly of Helsinki, Finland in 1964 and the modifications made by that assembly in Tokyo, Japan in 1975, in Venice, Italy in 1983, in Hong Kong in 1989 and the 54th General Assembly in Seoul Korea in 2008, where medical research is contemplated (Clinical Research). It will also be in accordance with what is specified by the General Health Law of Mexico, in the area of health research, in its article 17, considering the present study with a risk greater than the minimum. Likewise, the institutional norm of the IMSS for research of human beings will be followed. All participants will sign their written consent. Resources: Patients treated at the UMAE Hospital de Especialidades del CMNO. The protocol was approved with registration number R 2018 1001 079. Group Experience: The Advisor has the experience and scientific knowledge of the realization and publication of research studies (Level II and Level III of the SNI).

Study time: It will take place from October 2018 to June 2021.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of ischemic heart disease who will undergo surgery to CRC.
* Age 40 to 70 years.
* BMI from 18.5 to 29.9 kg / m2
* Stable renal function with a serum creatinine less than 1.5 mg / dl.
* Complete and signed informed consent.

Exclusion Criteria:

* Left ventricular ejection fraction <40%.
* Pre-existing disease such as: Renal impairment under substitute treatment (peritoneal dialysis or hemodialysis), Hepatic impairment, Human immunodeficiency syndrome, Viral liver disease (due to virus B and C).
* Patients with previous cardiac surgery.
* Emergency surgery or myocardial ischemia in progress.
* Known allergy to the supplement to be used in the study
* Alcohol abuse or drug use 1 month before surgery

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Troponin I | 24 hours
  Kit de Troponin-I ELISA, Biometrica, California, USA Evaluado a través de un analizador automático (ELx808 Absorbance Lector de microplacas; BioTek, Winooski, VT, EE. UU
Heat shock proteins 70 (HSP 70) | 24 hours
  Measurement in mononuclear cells in peripheral blood. Analyzed with Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD)
IL-6 IL-10 FNTα | 24 hours
  ELISA (KMI Diagnostics, Minneapolis, MN and Flanders, NJ). The results were obtained by spectrophotometry (Thermo Opsys MR Laboratory Systems, Chantily, VA).
CPK y CPK MB | 24 hours
  Analyzed with Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano del Seguro Social, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No